CLINICAL TRIAL: NCT06283784
Title: Double Blind, Randomized, Placebo Controlled Study To Evaluate The Efficacy of a Proprietary Mix of Live Probiotics in the Prophylaxis Of Diarrhea In Adult Patients Who Already Initiated An Oral Antibiotic Therapy
Brief Title: Study To Evaluate The Efficacy of a Proprietary Mix of Live Probiotics In The Prophylaxis Of Diarrhea In Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biofarma (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YOVIS Capsules
Record Dates: First submitted 2024-02-22; First posted 2024-02-28 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: This is a double blind, randomized, placebo-controlled study.
Who Masked: Participant, Investigator
Masking Description: YOVIS, the Investigational Food Supplement (IFS), is an oral formulation (capsules) containing definite mix of live probiotics. Placebo is an oral formulation of inert capsules. Placebo and YOVIS are identical in shape, size, colour and taste. Product test and placebo capsules will be indistinguishable.
  Investigational food supplement products will be packed in an individual way for each subject included in the investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yovis Capsules (Experimental): YOVIS, the Investigational Food Supplement (IFS), is an oral formulation (capsules) containing definite mix of live probiotics already marketed by Alfa-Sigma as food supplement since September 2017. it is administered to 50 patients 10 consecutive days (1 capsule once daily) with a drop of water, preferably without food.
  Interventions: Other: Yovis Capsules
- Placebo (Placebo Comparator): Placebo is an oral formulation of inert capsules. it is administered to 50 patients 10 consecutive days (1 capsule once daily) with a drop of water, preferably without food.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Yovis Capsules — Subjects will assume the active treatment for 10 consecutive days (1 capsule once daily) with a drop of water, preferably without food.
  Other Names: Probiothic
  Arms: Yovis Capsules
Other: Placebo — Subjects will assume the placebo treatment for 10 consecutive days (1 capsule once daily) with a drop of water, preferably without food.
  Arms: Placebo

SUMMARY:
This is a double blind, randomized, placebo-controlled study. One-hundred subjects are randomized to receive either YOVIS or placebo over a period of 10 days.

The purpose is to determinate the efficacy of the treatment in subjects treated with antibiotic therapy, by measuring occurrence of Antibiotic Associated Diarrhoea (AAD) from baseline to the end of the observation period (28±2 days)

DETAILED DESCRIPTION:
AAD is defined as clinically unexplained diarrhea that occurs in connection with antibiotic administration. Any antibiotic could potentially cause AAD, but broad-spectrum antibiotics that predominantly target anaerobes and are poorly absorbed, such as clindamycin, cephalosporins (cefixime and ceftriaxone), and amoxicillin-clavulanate, have a higher AAD incidence (Turck D, 2003). It has been reported that the highest rates of AAD in 650 pediatric cases were associated with amoxicillin/clavulanate (23%), penicillin A or M (11%) and erythromycin (16%).

In the present trial, adult population already under antibiotic therapy with ampicillin/amoxicillin, cephalosporins and clindamycin, will be selected, in order to capture the highest possible diarrhea events, with a limited number of subjects.

YOVIS, the Investigational Food Supplement (IFS), is an oral formulation (capsules) containing definite mix of live probiotics already marketed by Alfa-Sigma as food supplement since September 2017.

Placebo is an oral formulation of inert capsules. Placebo and YOVIS are identical in shape, size, colour and taste.

One-hundred (100) subjects will be randomized to receive either YOVIS or placebo (1:1) over a period of 10 days.

In case all inclusion/exclusion criteria are met, the subject will be randomized at the baseline visit to one of two masked trial treatments. Further phone contacts are scheduled on day 10±2 and day 21±2, a final visit at site is scheduled on day 28±2.

The primary objective of this study is to assess, versus placebo, the efficacy of a 10 days treatment with YOVIS in preventing the incidence of AAD in subjects under antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, personally signed and dated by the subject.
2. Subjects of both sexes between 18 and 65 years of age (limits included), with no limitation of race.
3. Patients being prescribed or having started an antibiotic therapy with ampicillin/amoxicillin, cephalosporins and clindamycin in the 48h preceding the screening.
4. Antibiotic therapy prescription with a lasting of at least 3 days but no more than 14 days.
5. Subject able to comprehend the full nature and purpose of the study, available to cooperate with the Investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

Inclusion criteria Subjects will be included in the study if they meet all the following criteria.

1. Written informed consent, personally signed and dated by the subject.
2. Subjects of both sexes between 18 and 65 years of age (limits included), with no limitation of race.
3. Patients being prescribed or having started an antibiotic therapy with ampicillin/amoxicillin, cephalosporins and clindamycin in the 48h preceding the screening.
4. Antibiotic therapy prescription with a lasting of at least 3 days but no more than 14 days.
5. Subject able to comprehend the full nature and purpose of the study, available to cooperate with the Investigator and to comply with the requirements of the entire study.

Exclusion Criteria

Subjects will be excluded if they meet any of the following criteria:

1. Pregnant or breast-feeding woman.
2. Known hypersensitivity or allergy to the active ingredients and/or to any component of the probiotic mix.
3. Subject with known food intolerance (eg. milk protein, gluten..)
4. Subject who has taken during the 2 weeks prior to inclusion, who is currently taking or plans to take other orally administered food supplements except the study product
5. Use of antidiarrhoeic drug is forbidden (maintenance of stable and regular treatment started more than 2 weeks before screening visit is allowed)
6. Active diarrhea at the time of the screening visit
7. Non controlled intestinal disease
8. Any antibiotic therapy in the 30 days preceding enrolment
9. Active participation in another clinical study
10. Subject with one or more psychiatric disturbances, such as: alcoholism, substance abuse or dependency disorder, bipolar disorder, schizophrenia, or other personality disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-05 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Efficacy of YOVIS in preventing the incidence of AADD in subjects under antibiotic therapy | 10 days - 21 days - 28 days
  The primary objective of this study is to assess, versus placebo, the efficacy of a 10 days treatment with YOVIS in preventing the incidence of AAD in subjects under antibiotic therapy. The incidence of diarrhea in the treatment group will be compared to placebo in the time frame of 28 days.

SECONDARY OUTCOMES:
Severity and duration of AAD | Time Frame: 28 days
  Cumulated duration of antibiotic-associated diarrhea (AAD) : number of days with diarrhea within the observation period
Severity and duration of AAD | Time Frame: 28 days
  Cumulative severity of antibiotic-associated diarrhea (AAD): sum of the values (obtained by transformation of Bristol stool form types) of all stools during days with diarrhea (transformation of Bristol scale types is defined: type 1 to 4 = 0; type 5 = 1; type 6 = 2 and type 7 = 3) diarrhea within the observation period
Evaluation of duration and severity of gastrointestinal symptoms | 28 days
  number of patients with gastrointestinal symptoms in the two groups
Evaluation of duration and severity of gastrointestinal symptoms | 28 days
  cumulative duration with symptoms in the two groups;
Evaluation of duration and severity of gastrointestinal symptoms | 28 days
  the cumulative severity of each symptom
Impact of bowel habits on QoL | 10-21-28 days
  assessed trough a 6-item questionnaire self-compiled by the subject at each visit. Quality of Life Questionnaire is compiled. 6 questions from minimum value of 0 (no impact) to 10 (maximum impact) on the quality of life
Effects of YOVIS, versus placebo, at each visit on the overall health status | 10-21-28 days
  assessed trough questions on the general well-being and through physical examination during visits. Questionnaire on the Gatrointestinal syntoms. each question minimum value is 0 (no pain at all) to 10 (maximum intensity of pain)
Assessment of acceptability, safety and satisfaction grade of YOVIS versus placebo | 10 days
  Patient satisfaction will be evaluated at the end of treatment. The clinician will ask the patient his satisfaction grade compared to her expectation, in a 5-point scale: Not at all Satisfied," "Partly Satisfied," "Satisfied," "More than Satisfied," "Very Satisfied," numbering 1 to 5 as an interval scale.
Global Patient's self-reported acceptance at the end of study | 28 days
  Global patient's acceptance to the treatment will be evaluated at the end of study visit, referred to the whole period, as bad, good, fair, excellent
Global acceptability (investigator) at the end of study | 28 days
  Global investigator acceptance to the treatment will be evaluated at the end of study visit, referred to the whole period, as bad, good, fair, excellent

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Agati, MD, Principal Investigator — General Practitioner
Locations (1):
- General Practitioner Ambulatory, Sanremo, Italy/Imperia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ashraf R, Shah NP. Immune system stimulation by probiotic microorganisms. Crit Rev Food Sci Nutr. 2014;54(7):938-56. doi: 10.1080/10408398.2011.619671. PMID 24499072
- [Result] Arvola T, Laiho K, Torkkeli S, Mykkanen H, Salminen S, Maunula L, Isolauri E. Prophylactic Lactobacillus GG reduces antibiotic-associated diarrhea in children with respiratory infections: a randomized study. Pediatrics. 1999 Nov;104(5):e64. doi: 10.1542/peds.104.5.e64. PMID 10545590
- [Result] Beaugerie L, Petit JC. Microbial-gut interactions in health and disease. Antibiotic-associated diarrhoea. Best Pract Res Clin Gastroenterol. 2004 Apr;18(2):337-52. doi: 10.1016/j.bpg.2003.10.002. PMID 15123074
- [Result] Chu W, Lu F, Zhu W, Kang C. Isolation and characterization of new potential probiotic bacteria based on quorum-sensing system. J Appl Microbiol. 2011 Jan;110(1):202-8. doi: 10.1111/j.1365-2672.2010.04872.x. Epub 2010 Oct 18. PMID 20955192
- [Result] Collado MC, Gonzalez A, Gonzalez R, Hernandez M, Ferrus MA, Sanz Y. Antimicrobial peptides are among the antagonistic metabolites produced by Bifidobacterium against Helicobacter pylori. Int J Antimicrob Agents. 2005 May;25(5):385-91. doi: 10.1016/j.ijantimicag.2005.01.017. PMID 15848292
- [Result] Cotter PD, Hill C, Ross RP. Bacteriocins: developing innate immunity for food. Nat Rev Microbiol. 2005 Oct;3(10):777-88. doi: 10.1038/nrmicro1273. PMID 16205711
- [Result] Hempel S, Newberry SJ, Maher AR, Wang Z, Miles JN, Shanman R, Johnsen B, Shekelle PG. Probiotics for the prevention and treatment of antibiotic-associated diarrhea: a systematic review and meta-analysis. JAMA. 2012 May 9;307(18):1959-69. doi: 10.1001/jama.2012.3507. PMID 22570464
- [Result] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Result] Lee YK, Puong KY, Ouwehand AC, Salminen S. Displacement of bacterial pathogens from mucus and Caco-2 cell surface by lactobacilli. J Med Microbiol. 2003 Oct;52(Pt 10):925-930. doi: 10.1099/jmm.0.05009-0. PMID 12972590
- [Result] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Result] Lui M, Gallo-Hershberg D, DeAngelis C. Development and validation of a patient-reported questionnaire assessing systemic therapy induced diarrhea in oncology patients. Health Qual Life Outcomes. 2017 Dec 22;15(1):249. doi: 10.1186/s12955-017-0794-6. PMID 29273046
- [Result] Lukasik J, Guo Q, Boulos L, Szajewska H, Johnston BC. Probiotics for the prevention of antibiotic-associated adverse events in children-A scoping review to inform development of a core outcome set. PLoS One. 2020 May 29;15(5):e0228824. doi: 10.1371/journal.pone.0228824. eCollection 2020. PMID 32469907
- [Result] Ritchie ML, Romanuk TN. A meta-analysis of probiotic efficacy for gastrointestinal diseases. PLoS One. 2012;7(4):e34938. doi: 10.1371/journal.pone.0034938. Epub 2012 Apr 18. PMID 22529959
- [Result] Servin AL. Antagonistic activities of lactobacilli and bifidobacteria against microbial pathogens. FEMS Microbiol Rev. 2004 Oct;28(4):405-40. doi: 10.1016/j.femsre.2004.01.003. PMID 15374659
- [Result] Turck D, Bernet JP, Marx J, Kempf H, Giard P, Walbaum O, Lacombe A, Rembert F, Toursel F, Bernasconi P, Gottrand F, McFarland LV, Bloch K. Incidence and risk factors of oral antibiotic-associated diarrhea in an outpatient pediatric population. J Pediatr Gastroenterol Nutr. 2003 Jul;37(1):22-6. doi: 10.1097/00005176-200307000-00004. PMID 12827001
- [Result] von Ossowski I, Reunanen J, Satokari R, Vesterlund S, Kankainen M, Huhtinen H, Tynkkynen S, Salminen S, de Vos WM, Palva A. Mucosal adhesion properties of the probiotic Lactobacillus rhamnosus GG SpaCBA and SpaFED pilin subunits. Appl Environ Microbiol. 2010 Apr;76(7):2049-57. doi: 10.1128/AEM.01958-09. Epub 2010 Jan 29. PMID 20118368